CLINICAL TRIAL: NCT03613272
Title: A Prospective Multicenter Comparative Study of the Curative Effect of Extended Thymectomy Performed Through the Subxiphoid VATS Approach With Double Elevation of the Sternum Versus Intercostal VATS Approach
Brief Title: The Curative Effect of Extended Thymectomy Performed Through Subxiphoid-right VATS Approach With Elevation of Sternum
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiang Fan (Other)
Responsible Party: Sponsor-Investigator, Jiang Fan, Chief physician, Tongji University
Organization: Tongji University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K18-137
Record Dates: First submitted 2018-07-07; First posted 2018-08-03 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Thymoma; Myasthenia Gravis; Mediastinal Tumor
Keywords: thymoma; thymectomy; Myasthenia Gravis; VATS; subxiphoid; elevation of the sternum; curative effect
MeSH Terms: conditions — Thymoma; Myasthenia Gravis; Mediastinal Neoplasms

STUDY DESIGN:
Intervention Model Description: This study is a prospective multicentre cohort study.The main study content is comparative study of the curative effect of extended thymectomy performed through the subxiphoid-right video-thoracoscopic approach with double elevation of the sternum versus intercostal video-thoracoscopic approach, divided into subxiphoid and intercostal groups. Communicating with the surgeon and patients who meet the inclusion criteria, decide whether to enter the subxiphoid or intercostal group. Subxiphoid group with subxiphoid-right video-thoracoscopic approach under double elevation of the sternum in extended thymectomy , intercostal group with traditional intercostal video-assisted thoracoscopic surgery in extended thymectomy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subxiphoid approach (Experimental): The patients in subxiphoid group will get subxiphoid approach extended thymectomy by VATS. Whole dissection was performed through a 4 to 7cm transverse subxiphoid incision, and a single 5-mm port was inserted into the right chest cavity for the video thoracoscope and subsequently for the chest tube. The sternum was elevated with two hooks connected to the sternal frame. The lower hook was inserted through the subxiphoid incision, and the superior hook was inserted percutaneously after the mediastinal tissue including the major mediastinal vessels was dissected from the inner surface of the sternum. The thymus and fatty tissue of the anterior mediastinum and the aorta-pulmonary window was completely removed.
  Interventions: Procedure: Subxiphoid approach extended thymectomy by VATS
- Intercostal approach (Experimental): The patients in intercostal group will get intercostal approach extended thymectomy by VATS.
  Interventions: Procedure: Intercostal approach extended thymectomy by VATS

INTERVENTIONS:
Procedure: Subxiphoid approach extended thymectomy by VATS — Extended thymectomy performed through the subxiphoid-right VATS approach with double elevation of the sternum
  Arms: Subxiphoid approach
Procedure: Intercostal approach extended thymectomy by VATS — Extended thymectomy performed through the traditional intercostal VATS approach
  Arms: Intercostal approach

SUMMARY:
Extended thymectomy is the main treatment for thymoma and other anterior mediastinal diseases. Video-assisted thoracic surgery(VATS) plays an important role in the surgery of extended thymectomy. Now, VATS thymectomy through intercostal approach has been the commonly used minimally invasive surgical procedure for thymus surgery and is applied worldwide. But the intercostal approach may cause residue of thymus tissue and chronic pain. In 2013, doctor Marcin Zielin´ski form Poland reported a new technique of minimally invasive extended thymectomy performed through the VATS approach with double elevation of the sternum. And their early results proved this technique is probably the least invasive and the most complete technique of VATS thymectomy with excellent cosmetic results. Until now, doctor Jiang Fan form Shanghai Pulmonary Hospital has performed 50 cases extended thymectomy through the subxiphoid approach with double elevation of the sternum by VATS. This study is designed to compare the curative effect between this new method and traditional intercostal VATS.

DETAILED DESCRIPTION:
This study is a prospective multicentre cohort study.The main study content is comparative study of the curative effect of extended thymectomy performed through the subxiphoid-right video-thoracoscopic approach with double elevation of the sternum versus intercostal video-thoracoscopic approach, divided into subxiphoid and intercostal groups. Communicating with the surgeon and patients who meet the inclusion criteria, decide whether to enter the subxiphoid or intercostal group. Subxiphoid group with subxiphoid-right video-thoracoscopic approach under double elevation of the sternum in extended thymectomy , intercostal group with traditional intercostal video-assisted thoracoscopic surgery in extended thymectomy. By collecting personal information of two groups of patients and the corresponding observation indicators to analyze whether the subxiphoid-right VATS approach with double elevation of the sternum is the least invasive and the most complete technique of VATS thymectomy.

ELIGIBILITY:
Inclusion Criteria:

1. MG with thymic hyperplasia, thymoma or other anterior mediastinum disease
2. Masaoka stagingⅠ-Ⅱ
3. Patients with normal cardio-pulmonary function before operation, BMI<30

Exclusion Criteria:

1. Unable to tolerate surgery
2. Masaoka staging Ⅲ-Ⅳ
3. Patients who have undergone previous surgery or radiotherapy
4. Myasthenia crisis
5. Chronic pain or using opioid analgesics before surgery
6. Preoperative mental disorders such as excessive anxiety
7. Patients who underwent previous mediastinal surgery or cardiac surgery
8. Patients with thoracic deformity

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Resection rate of thymus tissue | 1 month
  The thymus tissue resection rate was calculated by comparing the preoperative and postoperative CT images.
Acute Pain Score | 24 hours
  Visual analogue score (VAS-score) is to asses the development of acute pain after surgery. 11 point numeric rating scale of 0 represented "no pain"and a score of 10 represented "worst pain " in patients 24 hours after operation.
Life Quality of Patients | 6 months
  The EuroQol 5 Dimensions (EQ-5D) is used. EQ-5D is a standardized instrument developed by the EuroQol Group as a measure of health-related quality of life that can be used in a wide range of health conditions and treatments. EQ-5D includes self-reported quality of life, where 0 is the worst and 100 is the best imaginable health state.
Myasthenia Gravis remission rate | 1 year
  The Quantitative Myasthenia Gravis scale (QMG) is used. It includes 13 items, such as eyelid ptosis, diplopia, eyelid closure, speech, swallowing, vital capacity, lift, grip and lower extremity elevation. QMG can evaluate myasthenia, and total score of the scale is from 0 (no myasthenia) to 39 (the most severe myasthenia). If the difference between the two assessment scores is greater than 3.5, it is considered that the symptoms of myasthenia gravis relieved.
Disease-free survival | Up to 5 years
  From grouping to the recurrence of disease or the time of death due to disease progression.
Recurrence rate | Up to 5 years
  The rate of patients recurrence after surgery

SECONDARY OUTCOMES:
Mortality rate | Up to 5 years
  Death caused by operation or complications
Overall survival | Up to 5 years
  From grouping to any cause of death
Operation time | 1 week
  Time of the surgical operation
Length of stay | 1 month
  The time of the patients in hospital
Complication rate | 1 month
  The incidence rate of postoperative complications in the two groups
Chronic Pain Score | 6 months
  Visual analogue score (VAS-score) is to asses the development of chronic pain after surgery. 11 point numeric rating scale of 0 represented "no pain"and a score of 10 represented "worst pain " in patients 6 months after operation.

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - The Second Affiliated Hospital of Hainan Medical University, Haikou, Hainan
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - Shanxi Provincial Cancer Hospital, Taiyuan, Shanxi
  - Shaoxing Center Hospital, Shaoxing, Zhejiang
  - Taizhou Center Hospital (Taizhou Unoversity Hospital), Taizhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Zielinski M, Czajkowski W, Gwozdz P, Nabialek T, Szlubowski A, Pankowski J. Resection of thymomas with use of the new minimally-invasive technique of extended thymectomy performed through the subxiphoid-right video-thoracoscopic approach with double elevation of the sternum. Eur J Cardiothorac Surg. 2013 Aug;44(2):e113-9; discussion e119. doi: 10.1093/ejcts/ezt224. Epub 2013 Jun 12. PMID 23761413
- [Result] Zielinski M, Hauer L, Hauer J, Pankowski J, Nabialek T, Szlubowski A. Comparison of complete remission rates after 5 year follow-up of three different techniques of thymectomy for myasthenia gravis. Eur J Cardiothorac Surg. 2010 May;37(5):1137-43. doi: 10.1016/j.ejcts.2009.11.029. Epub 2010 Feb 8. PMID 20117014
- [Result] Friedant AJ, Handorf EA, Su S, Scott WJ. Minimally Invasive versus Open Thymectomy for Thymic Malignancies: Systematic Review and Meta-Analysis. J Thorac Oncol. 2016 Jan;11(1):30-8. doi: 10.1016/j.jtho.2015.08.004. PMID 26762737
- [Result] Takeo S, Sakada T, Yano T. Video-assisted extended thymectomy in patients with thymoma by lifting the sternum. Ann Thorac Surg. 2001 May;71(5):1721-3. doi: 10.1016/s0003-4975(00)02697-7. PMID 11383846
- [Result] Hess NR, Sarkaria IS, Pennathur A, Levy RM, Christie NA, Luketich JD. Minimally invasive versus open thymectomy: a systematic review of surgical techniques, patient demographics, and perioperative outcomes. Ann Cardiothorac Surg. 2016 Jan;5(1):1-9. doi: 10.3978/j.issn.2225-319X.2016.01.01. PMID 26904425